CLINICAL TRIAL: NCT01005745
Title: Lymphodepletion Plus Adoptive Cell Transfer With High Dose IL-2 in Patients With Metastatic Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15781
Record Dates: First submitted 2009-10-27; First posted 2009-11-02 (Estimated); Results first posted 2014-06-02 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Melanoma
Keywords: skin; adoptive cell therapy; tumor-infiltrating lymphocytes (TIL); lymphodepletion
MeSH Terms: conditions — Melanoma | interventions — Surgical Procedures, Operative; Lymphocyte Count; Cyclophosphamide; Adoptive Transfer; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TIL With High Dose IL-2 (Experimental): Day -7 and -6: Cyclophosphamide 60 mg/kg/day I.V. in 250 ml NS over approximately 2 hours. Mesna 20 mg/kg with D5W or NS at 125 ml/hour infused intravenously over 24 hours.
  Day -5 to Day -1: Fludarabine 25 mg/m^2 intravenous piggyback (IVPB0 daily over approximately 30 minutes for 5 days.
  Day 0: T cell infusion in 250-1000 ml NS over approximately 15-60 minutes depending on volume to be infused.
  Days 1-5: High dose IL-2, 720,000 IU/kg IV bolus (about 15 minutes) every 8-16 hours for up to 15 doses, beginning approximately 12-16 hours after T cell infusion.
  Interventions: Procedure: Surgery; Drug: Administration of Lymphodepletion; Other: Adoptive Cell Transfer; Drug: High Dose IL-2

INTERVENTIONS:
Procedure: Surgery — Surgery to remove a tumor for growth of TIL
  Other Names: Tumor Infiltrating Lymphocytes (TIL); T-cell; lymphocyte
Drug: Administration of Lymphodepletion — Lymphodepleting chemotherapy with cyclophosphamide and fludarabine to enhance T cell persistence and effectiveness in vivo
  Other Names: Cytoxan
Other: Adoptive Cell Transfer — T-cell infusion
Drug: High Dose IL-2 — Beginning approximately 12 - 16 hours after cell infusion.
  Other Names: Interleukin-2; Aldesleukin; Proleukin

SUMMARY:
The overall purpose of this research study is to find a better way to treat melanoma. This will be a single arm exploratory trial to evaluate prospectively the feasibility of, the toxicities of, and the persistence of TIL which can survive in vivo.

DETAILED DESCRIPTION:
Patients are being offered admission to this study to test the side effects of an investigational treatment prepared from special immune cells (T cells) specific for melanoma. A T-cell is a type of lymphocyte. Lymphocytes are a type of white blood cell that protect people from viral infections; help other cells fight bacterial and fungal infections; produce antibodies; fight cancers; and coordinate the activities of other cells in the immune system. These special immune cells will be taken from a sample of the patient's tumor tissue that will be surgically removed from their body and grown in the laboratory. They will then given back to the patient in their veins. These cells are called tumor infiltrating lymphocytes (TIL). We wish to study the side effects of TIL when they are given with two chemotherapy drugs to temporarily decrease the patient's own immune cells and a drug called Interleukin-2 (IL-2). The two chemotherapy drugs called fludarabine and cytoxan are used to greatly reduce the number of normal lymphocytes circulating in the patient's body, called lymphodepletion, so that there will be more "space" for the cancer fighting lymphocytes (T-cells) that will be infused in their veins. We wish to find out how often these cells can shrink or slow the growth of the patient's melanoma. We also wish to find out the effects of lymphodepletion followed by TIL and high dose IL-2 on the patient's immune system. The lymphodepletion followed by TIL and high dose IL-2 is experimental, and has not been proven to help treat melanoma.

The IL-2 has been approved by the Food and Drug Administration (FDA) for the treatment of metastatic melanoma that cannot be surgically removed. The chemotherapy drugs cytoxan and fludarabine used for lymphodepletion have been approved by the FDA, but not for the treatment of metastatic melanoma.

The combination of lymphodepletion followed by TIL and high dose IL-2 is not FDA approved but the FDA is permitting its use in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have unresectable metastatic stage IV melanoma or stage III in-transit or regional nodal disease.
* Residual measurable disease after resection of target lesion(s) for TIL growth
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 -1. ECOG performance status of 0-1 will be inferred if the patient's level of energy is ≥ 50% of baseline.
* Patients may be treatment-naïve or may have been previously treated for metastatic disease.
* Patients with a negative pregnancy test (urine or serum) must be documented at screening for women of childbearing potential (WOCBP).
* Adequate renal, hepatic and hematologic function, including creatinine of less than or equal to 1.7 gm/dL, total bilirubin less than or equal to 2.0 mg/dL, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dL, aspartic transaminase (AST) and alanine transaminase (ALT) of less than 3X institutional upper limit of normal (ULN), hemoglobin of 8 gm/dL or more, white blood count (WBC) of 3000 per mm³ and total granulocytes of 1000 per mm³ or more, and platelets of 100,000 per mm³ or more.
* Patients must have a positive screening Epstein-Barr virus (EBV) antibody titre on screening test.
* Patients with antibiotic allergies per se are not excluded; although the production of TIL for adoptive transfer includes antibiotics, extensive washing after harvest will minimize systemic exposure to antibiotics.
* Patients that had previously grown sterile, validated TIL under Good Manufacturing Practices (GMP) conditions on Moffitt Clinical trial protocol 15375 (Use of Excess Melanoma Tumor Specimens Not Required for Diagnostic Purposes for Validation of Tumor Infiltrating Lymphocyte [TIL] Growth Procedures) meeting the above criteria may be consented and enrolled in the current trial using the previously established TIL stored in the Cell therapies Core facility for up to 2 years.
* At screening, patients with ≤ 3 untreated central nervous system (CNS) metastases may be included provided none of the untreated lesions are > 1 cm in greatest dimension, and there is no peri-tumoral edema present on brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT] if MRI is contraindicated).
* At screening, patients with CNS metastases treated with either surgical resection and/or radiation therapy may be included. Patients may be included if the largest lesion is ≤ 1 cm, and there is no evidence of progressive CNS disease on brain imaging at least 28 days after treatment.
* At screening, patients may be included if the largest lesion is > 1 cm or > 3 in number, and there is no evidence of progressive CNS disease on brain imaging at least 90 days after treatment with surgery and/or radiation therapy.
* All laboratory and imaging studies must be completed and satisfactory within 30 days of signing the consent document.

Exclusion Criteria:

* Patients with active systemic infections requiring intravenous antibiotics, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system are excluded.
* Patients testing positive for human immunodeficiency virus (HIV) titre, Hepatitis B surface antigen, Hepatitis C antibody, Human T-lymphotropic virus (HTLV) I or II antibody, or both rapid plasma reagent (RPR) and fluorescein treponemal antibodies (FTA) positive are excluded.
* Patients who are pregnant or nursing
* Patients needing chronic, immunosuppressive systemic steroids
* Patients with autoimmune diseases that require immunosuppressive medications
* Presence of a significant psychiatric disease, which in the opinion of the principal investigator or his designee, would prevent adequate informed consent or render immunotherapy unsafe or contraindicated
* Patients with > 3 untreated CNS metastases or evidence of peri-tumoral edema will be excluded.
* Patients with ≤ 3 untreated CNS metastases but with at least one lesion >1 cm or peri-tumoral edema will be excluded.
* Patients with treated CNS metastases > 1 cm or > 3 in number will be excluded if there is evidence of progressive CNS disease on brain imaging at least 90 days after treatment with surgery and/or radiation therapy.
* Inability to comprehend and give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-10-20 (Actual); Primary Completion 2014-01-31 (Actual); Study Completion 2025-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amod Sarnaik, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Moffitt Cancer Center from October 20, 2009 until November 15, 2012.
Groups:
- TIL With High Dose IL-2: Day -7 and -6: Cyclophosphamide 60 mg/kg/day I.V. in 250 ml NS over approximately 2 hours. Mesna 20 mg/kg with D5W or NS at 125 ml/hour infused intravenously over 24 hours.
  Day -5 to Day -1: Fludarabine 25 mg/m^2 intravenous piggyback (IVPB0 daily over approximately 30 minutes for 5 days.
  Day 0: T cell infusion in 250-1000 ml NS over approximately 15-60 minutes depending on volume to be infused.
  Days 1-5: High dose IL-2, 720,000 IU/kg IV bolus (about 15 minutes) every 8-16 hours for up to 15 doses, beginning approximately 12-16 hours after T cell infusion.
  Surgery: Surgery to remove a tumor for growth of TIL
  Administration of Lymphodepletion: Lymphodepleting chemotherapy with cyclophosphamide and fludarabine to enhance T cell persistence and effectiveness in vivo
  Adoptive Cell Transfer: T-cell infusion
  High Dose IL-2: Beginning approximately 12 - 16 hours after cell infusion.
Period: Overall Study
Arm/Group | TIL With High Dose IL-2
Started | 19
Completed | 13
Not Completed | 6
Not completed — No TIL growth | 1
Not completed — Disease progressed during TIL growth | 3
Not completed — Death prior to treatment | 1
Not completed — Inappropriate antidiuretic hormone | 1

BASELINE CHARACTERISTICS:
Population: All 19 participants accrued are listed for baseline, Primary Outcome Measure and Adverse Events. All 13 participants who completed treatment are listed for analysis of Secondary Outcome Measure.
Arm/Group | TIL With High Dose IL-2
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 46.5 [25 to 68]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Tumor Infiltrating Lymphocytes (TIL) Growth
Description: Feasibility was the primary endpoint of this trial, defined as a patient who can grow and expand T-cells: Number of participants with fragments cultured; Number of participants with fragments that reached a final count of 20e6 cells within 5 weeks of culture; Number of participants with fragments that reached a final count of 20e6 cells within 5 weeks of culture and were cocultured with autologous or human leukocyte antigen (HLA)-matched tumor cells for interferon(IFN)-γ production; Number of participants with fragments that produced IFN-γ in response to autologous or HLA-matched tumor cells.
Time Frame: 192 Days Post Surgical Resection
Population: All participants
Measure: Number; unit: participants
Arm/Group | TIL With High Dose IL-2
Number analyzed (Participants) | 19
participants
  Participants with fragments cultured | 19
  Participants with fragments grown | 14
  Participants with fragments tested | 14
  Participants with IFN-γ positive fragments | 13

2. Secondary Outcome: Number of Participants With Objective Response (OR)
Description: OR is defined as the patient being alive at Day 70 and tumor size evaluated using the Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria to be a complete response or partial response. Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. Evaluations were made by computed tomography (CT) scan approximately 6 to 8 weeks after the cell infusion, or CT scan approximately 10 weeks after the cell infusion, or by clinical evaluation during the first 70 days.
Time Frame: Average of 10 Months Follow-up
Population: All participants who completed treatment
Measure: Number; unit: participants
Arm/Group | TIL With High Dose IL-2
Number analyzed (Participants) | 13
participants
  Partial Response (PR) | 3
  Complete Response (CR) | 2
  Complete Response (PR + CR) | 5

ADVERSE EVENTS:
Time Frame: 3 years
Description: All participants
Arm/Group | TIL With High Dose IL-2
Serious Adverse Events (participants affected / at risk) | 7/19
Other Adverse Events (participants affected / at risk) | 14/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TIL With High Dose IL-2 (N=19)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Uveitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Blood antidiuretic hormone abnormal (Investigations) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other - basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Invasive squamous cell (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other - pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TIL With High Dose IL-2 (N=19)
Fatigue (General disorders) | 14 (32)
Chills (General disorders) | 13 (17)
Edema - limbs (General disorders) | 5 (9)
General disorders and administration site - Other (Gastrointestinal disorders) | 3 (4)
Pain (General disorders) | 3 (3)
Fever (General disorders) | 2 (3)
Edema - trunk (General disorders) | 1 (1)
Platelet count decreased (Investigations) | 13 (84)
White blood cell decreased (Investigations) | 13 (52)
Alkaline phosphatase increased (Investigations) | 10 (19)
Blood bilirubin increased (Investigations) | 10 (23)
Alanine aminotransferase increased (Investigations) | 8 (11)
Creatinine increased (Investigations) | 8 (13)
Lymphocyte count decreased (Investigations) | 8 (27)
Aspartate aminotransferase increased (Investigations) | 7 (12)
Neutrophil count decreased (Investigations) | 7 (22)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Blood antidiuretic hormone abnormal (Investigations) | 1 (1)
Investigations - Other (Investigations) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 13 (29)
Hypocalcemia (Metabolism and nutrition disorders) | 12 (43)
Hypophosphatemia (Metabolism and nutrition disorders) | 12 (23)
Anorexia (Metabolism and nutrition disorders) | 10 (13)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (42)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (25)
Hypomagnesemia (Metabolism and nutrition disorders) | 9 (17)
Hypokalemia (Metabolism and nutrition disorders) | 4 (7)
Hypermagnesemia (Metabolism and nutrition disorders) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 13 (71)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (9)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 7 (24)
Sinus tachycardia (Cardiac disorders) | 10 (14)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Cardiac disorders - Other (Cardiac disorders) | 3 (4)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 13 (19)
Vomiting (Gastrointestinal disorders) | 10 (15)
Diarrhea (Gastrointestinal disorders) | 9 (12)
Constipation (Gastrointestinal disorders) | 3 (5)
Mucositis oral (Gastrointestinal disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 9 (9)
Capillary leak syndrome (Vascular disorders) | 4 (4)
Vascular disorders - Other (Vascular disorders) | 4 (5)
Flushing (Vascular disorders) | 2 (2)
Hot flashes (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (7)
Dizziness (Nervous system disorders) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Sinus pain (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Confusion (Psychiatric disorders) | 4 (6)
Anxiety (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 2 (2)
Delirium (Psychiatric disorders) | 1 (3)
Acute kidney injury (Renal and urinary disorders) | 3 (8)
Urinary retention (Renal and urinary disorders) | 3 (3)
Proteinuria (Renal and urinary disorders) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (3)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (2)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (2)
Urine discoloration (Renal and urinary disorders) | 1 (2)
Cytokine release syndrome (Immune system disorders) | 3 (3)
Immune system disorders - Other (Immune system disorders) | 3 (4)
Blurred vision (Eye disorders) | 2 (2)
Flashing lights (Eye disorders) | 2 (3)
Cataract (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Uveitis (Eye disorders) | 1 (1)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes